CLINICAL TRIAL: NCT00308763
Title: Clinical Trial of Two Medications on Smoking Cessation
Brief Title: Nicotine Patch and Bupropion to Reduce Smoking Rates in Younger, Low-Income, and Minority Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 376; R01HL066025 (NIH); R01HL066025-05 (NIH)
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Nicotine patch plus placebo sustained-release bupropion
  Interventions: Drug: Nicotine Patch
- 2 (Active Comparator): Placebo nicotine patch plus sustained-release bupropion
  Interventions: Drug: Sustained Release Bupropion
- 3 (Active Comparator): Nicotine patch plus sustained-release bupropion
  Interventions: Drug: Nicotine Patch; Drug: Sustained Release Bupropion

INTERVENTIONS:
Drug: Nicotine Patch — After determining that it is appropriate to dispense study medication to a participant, the dosing regimen will be determined. Participants who report smoking more than 20 cigarettes each day will be initially placed on the 21 mg patch; participants who report smoking 10 - 19 cigarettes each day will be initially placed on the 14 mg patch; participants who report smoking 5 - 9 cigarettes will be initially placed on the 7 mg patch.
  If a participant is initially placed on the 21 mg patch, the following dosing schedule will occur: 21 mg patch for 4 weeks, 14 mg patch for 4 weeks, 7 mg patch for 2 weeks, and then off. If a participant is initially placed on the 14 mg patch, the following dosing schedule will occur: 14 mg patch for 6 weeks, 7 mg patch for 4 weeks, and then off. If a participant is initially placed on the 7 mg patch, the following dosing schedule will occur: 7 mg patch for 10 weeks, and then off.
  Arms: 1; 3
Drug: Sustained Release Bupropion — Participants will receive the sustained-release bupropion 150 mg tablet in the morning for four days. If this dose is well-tolerated, then the dose will be increased to a 150 mg tablet twice daily, with at least 8 hours between the two doses. The sustained-release bupropion medication will begin at the randomization visit (RV) which is approximately one week before the quit date. At the RV, the participant should be dispensed enough of the 150 mg tablets of the sustained-release bupropion or placebo to return for the first follow-up visit with instructions on use. Participants will be evaluated by telephone on their quit date approximately one week after the RV to assess safety. We will discontinue the sustained-release bupropion at the second follow-up visit, at which time participants will have received sustained-release bupropion for approximately 11 weeks.
  Arms: 2; 3

SUMMARY:
Nicotine addiction is a serious health problem in the United States; 46 million people smoke cigarettes, and 70% of those are trying to quit. The nicotine patch and bupropion, a medication used to reduce nicotine cravings, are two commonly used smoking cessation aids. Both have been shown to reduce smoking rates, however, the effectiveness of combining the two treatments has not been widely examined. This study will evaluate the effectiveness of the nicotine patch combined with bupropion at reducing smoking rates among younger, low-income, and minority individuals.

DETAILED DESCRIPTION:
Cigarette smoking poses a serious but preventable health risk. The negative health effects of smoking are well-known, but the prevalence of cigarette smoking remains high in the United States, particularly among younger people, people of lower socioeconomic status, and minority groups. Nicotine replacement therapy, commonly known as the nicotine patch, has been proven to be an effective treatment for reducing nicotine use. The nicotine patch provides a measured dose of nicotine through the skin. By gradually lowering nicotine doses over a period of time, individuals experience fewer nicotine cravings; the ultimate goal is to stop using nicotine. Bupropion, a medication commonly used to treat depression, is also used as a smoking cessation tool. It helps to control nicotine cravings. The majority of studies on the nicotine patch and bupropion have been performed on older, white, middle-class individuals; more research is needed to confirm the benefit of these treatments in younger, low-income, and minority populations. While both the nicotine patch and bupropion appear to be individually effective as smoking cessation aids, little is known on the possible effectiveness of combining the two treatments. Because of the high relapse rates in low-income and minority individuals, the combination of the nicotine patch with bupropion may be particularly effective at reducing relapse rates in these individuals. The purpose of this study is to evaluate the effectiveness of the nicotine patch and bupropion at reducing smoking rates in younger, low-income, and minority individuals.

This 1-year study will enroll younger, low-income, and minority individuals who smoke. Participants will be randomly assigned to one of the following three groups: 1) nicotine patch plus placebo sustained-release bupropion; 2) placebo nicotine patch plus sustained-release bupropion; or 3) nicotine patch plus sustained-release bupropion. At study entry, participants will complete standardized psychological questionnaires to assess depression levels and will undergo a physical exam and blood testing. Study visits will take place at Weeks 5 and 11, Month 6, and Year 1. At each visit, questionnaires will be completed, and smoking cessation rates will be assessed by self-report and verified by saliva and exhaled carbon monoxide testing. In addition, all participants will take part in a standardized behavioral smoking cessation program.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* In a lower socioeconomic group, defined as below median income in the study county
* Smokes more than 5 cigarettes each day for at least 6 months prior to study entry, as determined by self-report

Exclusion Criteria:

* History of a seizure disorder, brain tumor, or severe head trauma
* History of substance abuse, including alcohol use in excess of 14 drinks a week
* History of anorexia or bulimia
* History of cerebral, coronary, or peripheral vascular disease
* History of serious heart arrhythmia
* Presence of an unstable psychiatric illness
* Current use of a psychotropic medication, including antidepressant medications
* History of peptic ulcer disease or currently taking an H2 blocker (e.g., cimetidine)
* History of kidney disease, defined as creatinine levels greater than 1.5 times the upper limit of normal
* History of liver disease, defined as serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase(SGPT) levels greater than twice the upper limit of normal
* History of uncontrolled hyperthyroidism or pheochromocytoma
* History of atopic or eczematous dermatitis
* Current use of a medication that cannot be discontinued and may interfere with study procedures or may increase the risk of side effects (e.g., nicotine gum, nicotine nasal spray, theophylline, systemic steroids, levodopa)
* History of an allergic reaction to the nicotine patch or bupropion
* History of diabetes treated with an oral agent or insulin
* Uncontrolled high blood pressure, defined as blood pressure level greater than 140/90 mm Hg
* Severe uncontrolled asthma, bronchitis, or emphysema
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 594 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rates (measured by self-report, saliva test, and exhaled carbon monoxide test) | Measured at 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Karen C. Johnson, MD, MPH, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center / Department of Preventive Medicine, Memphis, Tennessee, United States

REFERENCES:
- [Result] Badrun F, Tolley B, Johnson KC. Smoking Cessation Interventions and Their Effects on Mood and Quit Pattern. In preparation 2014.